CLINICAL TRIAL: NCT05918965
Title: Effects of Transcutaneous Electrical Neurostimulation on Female Patients With Long COVID - a Pilot Study
Brief Title: Vagus Stimulation in Female Long COVID Patients.
Acronym: Vagus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Richard Crevenna, Head of Physical Medicine, Rehabilitation and Occupational Medicine, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1779/2022
Record Dates: First submitted 2023-06-20; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Vagus Nerve Diseases; Long COVID; Long Covid19; Post-COVID-19 Syndrome; Post-COVID Syndrome; Post COVID-19 Condition; Post COVID Condition
Keywords: auricular transcutaneous electrical vagal nerve stimulation; TENS
MeSH Terms: conditions — Vagus Nerve Diseases; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vagus Nerve Stimulation with 10 Hertz (Active Comparator): Twelve weeks home therapy with transcutaneous electrical neurostimulation (TENSeco®, CE197, Schwa-Medico Gmbh), transcutaneous 2-channel nerve stimulator.
  Matching ear electrode 3 DTS.
  * Stimulation frequency: 10 Hertz
  * Intensity: sensitive threshold; clearly perceptible, but pleasant
  * Form of stimulation: biphasic
  * Duration: 30 min
  * Position: left ear
  * Frequency: daily, in the evening, when all daily activities are done
  Interventions: Device: transcutaneous electrical vagal neurostimulation
- Vagus Nerve Stimulation with 25 Hertz (Active Comparator): Twelve weeks home therapy with transcutaneous electrical neurostimulation (TENSeco®, CE197, Schwa-Medico Gmbh), transcutaneous 2-channel nerve stimulator.
  Matching ear electrode 3 DTS.
  * Stimulation frequency: 25 Hertz
  * Intensity: sensitive threshold; clearly perceptible, but pleasant
  * Form of stimulation: biphasic
  * Duration: 30 min
  * Position: left ear
  * Frequency: daily, in the evening, when all daily activities are done
  Interventions: Device: transcutaneous electrical vagal neurostimulation
- Vagus Nerve Stimulation with 2 Hertz (Experimental): Twelve weeks home therapy with transcutaneous electrical neurostimulation (TENSeco®, CE197, Schwa-Medico Gmbh), transcutaneous 2-channel nerve stimulator.
  Matching ear electrode 3 DTS.
  * Stimulation frequency: 2 Hertz
  * Intensity: sensitive threshold; clearly perceptible, but pleasant
  * Form of stimulation: biphasic
  * Duration: 30 min
  * Position: left ear
  * Frequency: daily, in the evening, when all daily activities are done
  Interventions: Device: transcutaneous electrical vagal neurostimulation

INTERVENTIONS:
Device: transcutaneous electrical vagal neurostimulation — daily for 12 weeks

SUMMARY:
The aim of the present pilot study is to investigate the acceptance, feasibility and implementation of the vagus nerv stimulation in Long COVID patients. Additionally, the effects on parameters of the autonomic nervous system as well as on symptoms of Long COVID will be described in a pre/post comparison.

For this purpose, a total of 45 female Long COVID patients will participate in the randomized controlled pilot study. Patients will perform auricular vagus stimulation daily for 12 weeks. The patient collective will be randomized into three groups (A: 10 hertz, B: 25 hertz, C: 2 hertz=control group).

If appropriate results are obtained, further adequately powered intervention studies are planned.

DETAILED DESCRIPTION:
Patients start on day 0, when the first assessment takes place. This consists of a medical diagnostic interview and sociodemographic, anthropometric, medical and functional data are collected (for a detailed description, see chapter 5. Statistics). Subsequently, the patients fill out the given questionnaires (paper/pencil version), which are then evaluated. Subsequently, the test persons are trained by a doctor how the electrical stimulation works with a demo device. Finally, the device is taken over by the company Schwa-Medico. The whole first assessment lasts about 2 hours and always takes place from 8 a.m. at constant room temperature (22-23 C°).

The outcome parameters are recorded before the start of the vagus nerve stimulation (T0), during the treatment after 4 weeks (T0+4Wo) and after a total of 12 weeks (T0+12Wo) after the end of the therapy. Which assessments are collected at the different time points is listed in the biometry section. The assessments are performed by physicians of the Department of Physical Medicine, Rehabilitation and Occupational Medicine. All assessments take place at relatively the same time, at constant room temperature (22-23 C°). The patients have to appear fasting.

T0: Medical history, examination, randomization, pre-tests, enrollment. T0+4Wo: Intermediate examination T0+12Wo: final examination, post-tests, return of device

This pilot study investigates the acceptability, feasibility, and implementation of the VNS measure in Long COVID patients. In addition, effects on autonomic nervous system parameters (heart rate, blood pressure, rate pressure product, heart rate variability = HRV, cortisol in saliva), on symptoms fatigue, dyspnea as well as health-related quality of life (HRQOL) are described:

Time points: T0, T0+4wk, T0+12wk.

Parameters - collected at relatively the same time each day, at constant room temperature (22-23 C°):

* Documentation of blood pressure and pulse rate: by means of Boso Medicus (Bosch + Sohn GmbH u. Co. KG, Jungingen, Germany), calculation of the so-called "rate pressure-product" (syst. blood pressure x heart rate)
* Heart rate variability
* Salivary cortisol
* Fatigue: Brief Fatigue Inventory (BFI)
* Health-related quality of life (HRQOL): SF-36 (short form) questionnaire instrument
* Dyspnea: Modified Borg Scale
* Sleep: Insomnia Severity Index (ISI)

ELIGIBILITY:
Inclusion Criteria:

* Female patients with Long COVID (history, physical examination, findings)
* age 18-70 years
* signed informed consent

Exclusion Criteria:

* Hearing aid implants (cochlear implants)
* surgical transection of the vagus nerve
* Malignancies
* autoimmune diseases
* orthopedic diseases
* rheumatological diseases
* neurological diseases
* postoperative, fresh injuries to the ear
* febrile diseases
* inflammations
* psychiatric diseases
* pacemakers
* implanted cardioverter and defibrillators (ICDs)
* seizure disorders
* Meniere's disease
* negative experience with electrotherapy
* insufficient knowledge of the German language

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — More women are affected by Long Covid, also the homogeneity is granted in a small study population.
Enrollment: 45 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 3 times for 12 weeks
  20-minute documentation of the heart rate variability with a 24-hour-elektrocardiography

SECONDARY OUTCOMES:
blood pressure and pulse | 3 times for 12 weeks
  via Boso Medicus plus their mutiplication for the rate-pressure-product
Saliva cortisol | 3 times for 12 weeks
  in the morning until the latest 10am
Questionnaire Brief Fatigue Inventory (BFI) | 3 times for 12 weeks
  Fatigue evaluation
Questionnaire Short form (SF)-36 | 3 times for 12 weeks
  Health related quality of life evaluation
Questionnaire Borg-Scale | 3 times for 12 weeks
  Dyspnea evaluation
Questionnaire Insomnia Severity Index (ISI) | 3 times for 12 weeks
  Sleep evaluation
Post-COVID-19 Functional Status scale (PCFS) | 3 times for 12 weeks
  Grade 0-4

CONTACTS AND LOCATIONS:
Overall Officials: Richard Crevenna, M.D., Principal Investigator — PMR&O
Locations (1):
- Department of Physical Medicine, Rehabilitation and Occupational Medicine, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raveendran AV, Jayadevan R, Sashidharan S. Long COVID: An overview. Diabetes Metab Syndr. 2021 May-Jun;15(3):869-875. doi: 10.1016/j.dsx.2021.04.007. Epub 2021 Apr 20. PMID 33892403
- [Background] Shah W, Hillman T, Playford ED, Hishmeh L. Managing the long term effects of covid-19: summary of NICE, SIGN, and RCGP rapid guideline. BMJ. 2021 Jan 22;372:n136. doi: 10.1136/bmj.n136. No abstract available. PMID 33483331
- [Background] Sylvester SV, Rusu R, Chan B, Bellows M, O'Keefe C, Nicholson S. Sex differences in sequelae from COVID-19 infection and in long COVID syndrome: a review. Curr Med Res Opin. 2022 Aug;38(8):1391-1399. doi: 10.1080/03007995.2022.2081454. Epub 2022 Jun 20. PMID 35726132
- [Background] Dani M, Dirksen A, Taraborrelli P, Torocastro M, Panagopoulos D, Sutton R, Lim PB. Autonomic dysfunction in 'long COVID': rationale, physiology and management strategies. Clin Med (Lond). 2021 Jan;21(1):e63-e67. doi: 10.7861/clinmed.2020-0896. Epub 2020 Nov 26. PMID 33243837
- [Background] Fudim M, Qadri YJ, Ghadimi K, MacLeod DB, Molinger J, Piccini JP, Whittle J, Wischmeyer PE, Patel MR, Ulloa L. Implications for Neuromodulation Therapy to Control Inflammation and Related Organ Dysfunction in COVID-19. J Cardiovasc Transl Res. 2020 Dec;13(6):894-899. doi: 10.1007/s12265-020-10031-6. Epub 2020 May 26. PMID 32458400